CLINICAL TRIAL: NCT06305676
Title: Biomarker Approach to Screening for the Early Detection of HPV-related Oropharyngeal Cancer (BASH OPC)
Acronym: BASH OPC
Status: Recruiting | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: MCC-23073
Record Dates: First submitted 2024-03-06; First posted 2024-03-12 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Oropharyngeal Cancer; HPV-Related Carcinoma
Keywords: Oropharyngeal Cancer; Early Detection; Screening
MeSH Terms: conditions — Oropharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case Group: Case group will consist of early and late disease pre-treatment Oropharyngeal Cancer cases.
  Interventions: Diagnostic Test: combined HPV 16 DNA and host gene methylation oral biomarker panel
- Control Group: Controls will be enrolled from members of the catchment area to ensure geographic comparability of cases and controls. Controls will be matched by sex, age, race/ethnicity, and tobacco use.
  Interventions: Diagnostic Test: combined HPV 16 DNA and host gene methylation oral biomarker panel

INTERVENTIONS:
Diagnostic Test: combined HPV 16 DNA and host gene methylation oral biomarker panel — DNA Methylation Profiling

SUMMARY:
Investigators seek to determine the sensitivity and specificity of a combined HPV 16 DNA and host gene methylation oral biomarker panel to distinguish early Oropharyngeal Cancer (OPC) cases from controls among 100 early and 100 late disease pre-treatment OPC cases, and 200 controls matched by sex, age, race/ethnicity, and tobacco use collected from the Moffitt Cancer Center (Moffitt) and the University of Pittsburgh Medical Center Hillman Cancer Center (Pittsburgh).

ELIGIBILITY:
Inclusion Criteria:

Cases:

* Aged at least 18 years
* Newly diagnosed primary tumor, histologically confirmed squamous cell carcinoma of the oropharynx (stages I-IV)
* Has not received treatment (surgery, chemotherapy, radiation, or immunotherapy) within the previous four weeks
* Provided written informed consent under Moffitt Cancer Center (MCC) 17716 biomarker/biobanking study or is identified and enrolled at the University of Pittsburgh Medical Center Hillman Cancer Center
* Aged at least 35 years
* Have no previous diagnosis of HNC or HPV-related cancer
* Fully understands study procedures
* Voluntarily agrees to participate by giving written informed consent under Moffitt Cancer Center (MCC) 17716 biomarker/biobanking study or is enrolled at the University of Pittsburgh Medical Center Hillman Cancer Center

Exclusion Criteria:

* Not meeting all of the above inclusion criteria for either the case or control group

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 100 early and 100 late disease pre-treatment Oropharyngeal Cancer cases, and 200 controls matched by sex, age, race/ethnicity, and tobacco use collected from the Moffitt Cancer Center (Moffitt) and the University of Pittsburgh Medical Center Hillman Cancer Center (Pittsburgh).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Sensitivity | Up to 60 months
  A 95% one-sided confidence interval using the Wilson method will be obtained for sensitivity for the early Oropharyngeal Cancer cases and late Oropharyngeal Cancer cases.
Diagnostic Specificity | Up to 60 months
  A 95% one-sided confidence interval using the Wilson method will be obtained for Specificity based on the control patients.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Giuliano, PhD, Principal Investigator — Moffitt Cancer Center; Antonio Amelio, PhD, Principal Investigator — Moffitt Cancer Center
Locations (2):
- United States (2):
  - Moffitt Cancer Center, Tampa, Florida
  - University of Pittsburgh Medical Center (UPMC) Hillman Cancer Center, Pittsburgh, Pennsylvania

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials Website — http://www.moffitt.org/clinical-trials-research/clinical-trials/